CLINICAL TRIAL: NCT02708511
Title: 64Cu-DOTA-B-Fab as A PET Tracer for Evaluating CA6 Expression in Tumors: A First in Human Study
Brief Title: Copper Cu 64-DOTA-B-Fab PET/CT in Imaging Patients With Ovarian and Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sanjiv Sam Gambhir (Other)
Responsible Party: Sponsor-Investigator, Sanjiv Sam Gambhir, Virginia and D.K. Ludwig Professor for Clinical Investigation in Cancer Research, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GYNOVA0033; NCI-2015-00767 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 32991; GYNOVA0033 (Other: Stanford Cancer Institute); IRB-32991 (Other: Stanford IRB)
Record Dates: First submitted 2015-11-16; First posted 2016-03-15 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Ovarian Carcinoma; Breast Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms | interventions — Tomography, X-Ray Computed; Tomography; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Diagnostic (Cu 64 DOTA-B-Fab) (Experimental): Patients receive copper Cu 64-DOTA-B-Fab IV followed by PET/CT 60 minutes post-injection and 24 hours post-injection
  Interventions: Diagnostic Test: Computed Tomography; Drug: Copper Cu 64-DOTA B-Fab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Diagnostic Test: Positron Emission Tomography

INTERVENTIONS:
Diagnostic Test: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Drug: Copper Cu 64-DOTA B-Fab — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Diagnostic Test: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot clinical trial studies copper Cu 64-DOTA-B-Fab positron emission tomography (PET)/computed tomography (CT) in imaging patients with ovarian and breast cancer. Cancer antigen (CA)6 is an antigen (substance) found on the surface of several types of cancer cells such as cancer of the ovary and breast. Diagnostic procedures, such as copper Cu 64-DOTA-B-Fab PET/CT, may help identify CA6 positive tumors and allow doctors to plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dosimetry of 64Cu-DOTA B-Fab (copper Cu 64-DOTA-B-Fab).

SECONDARY OBJECTIVES:

I. To evaluate the safety of 64Cu-DOTA B-Fab single administration.

II. To evaluate the ability of 64Cu-DOTA B-Fab to detect CA6-positive ovarian and breast cancer lesions.

III. To compare PET results with the immunohistochemistry (IHC) analysis of the excised tumor samples.

OUTLINE:

Patients receive copper Cu 64-DOTA-B-Fab intravenously (IV) followed by PET/CT 60 minutes post-injection and 24 hours post-injection

After completion of study, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

Ovarian Cancer Participants

1. Patient is ≥ 18 years old at the time of the drug administration
2. Participant has suspected or biopsy proven ovarian cancer and is scheduled to undergo surgical excision of the cancerous lesion(s) OR Participant has biopsy proven ovarian cancer but is not a surgical candidate
3. Ability to understand and the willingness to sign a written informed consent document.
4. Patient is able to remain still for duration of each imaging procedure

Breast Cancer Participants

1. Patient is ≥ 18 years old at the time of the drug administration
2. Participant has biopsy proven breast cancer and may or may not undergo surgical excision of the cancerous lesion(s)
3. Ability to understand and the willingness to sign a written informed consent document.
4. Patient is able to remain still for duration of each imaging procedure

Exclusion Criteria:

Ovarian Cancer Participants

1. Patient is pregnant or breast-feeding
2. Patients with contraindications for PET/CT or who cannot complete a PET/CT scan or other study procedures.
3. Patients with serious uncontrolled concurrent medical illness that would limit compliance with study requirements
4. Patients participating in other research imaging protocols will be excluded from this study.

Breast Cancer Participants

1. Patient is pregnant or breast-feeding
2. Patients with contraindications for PET/CT or who cannot complete a PET/CT scan or other study procedures.
3. Patients with serious uncontrolled concurrent medical illness that would limit compliance with study requirements
4. Patients participating in other research imaging protocols will be excluded from this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-08; Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Biodistribution of copper Cu 64 DOTA-B-Fab | 24 hours
  Determined from serial imaging correlated with blood and urine samples.
Dosimetry of copper Cu 64 DOTA-B-Fab | 120 minutes post-injection
  Determined from serial imaging correlated with blood and urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Gambhir, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States